CLINICAL TRIAL: NCT00862862
Title: Evaluation of Pharmacodynamic Target Attainment With Vancomycin Treatment of Infections Due to Staphylococcus Aureus
Brief Title: Evaluation of Vancomycin Treatment of Infections Due to Staphylococcus Aureus
Status: Terminated | Type: Observational
Why Stopped: lack of enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0002-09-FB
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Staphylococcus Aureus
Keywords: infection; staphylococcus aureus; vancomycin; pharmacodynammics
MeSH Terms: conditions — Staphylococcal Infections; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: The objective of the study is to evaluate the ability of current vancomycin dosing strategies to attain the pharmacodynamic target of an area under the curve (AUC) to minimum inhibitory concentration (MIC) ratio greater than 400:1 for patients with a suspected or documented Staphylococcus aureus infection.

Primary Outcome: The primary outcome is the percentage of vancomycin dosing regimens that achieve AUC:MIC ratio > 400 on the first occurrence of vancomycin use in patients with a suspected or documented S. aureus infection at The Nebraska Medical Center.

Secondary Outcomes:

1. To assess the probability that vancomycin AUC:MIC ratios obtained from The Nebraska Medical Center patients exceed a therapeutic threshold using S. aureus MICs from isolates obtained from The Nebraska Medical Center.
2. Using MIC data from the TRUST Study database (large national surveillance database) and the vancomycin AUC data obtained from TNMC patients, perform a Monte Carlo analysis that will assess the probability of achieving a therapeutic vancomycin threshold with a large number of isolates.

DETAILED DESCRIPTION:
Study Design: This is a prospective cohort study with a retrospective chart review component.

Inclusion and Exclusion Criteria: Inpatients of The Nebraska Medical Center will be included if they are 19 years of age or older, prescribed intravenous vancomycin therapy with a dosing interval of 24 hours or less, and therapy is continued for at least 3 doses or five half lives. Exclusion criteria consists of an estimated creatinine clearance less than 30 ml/min, concurrent use of dialysis, and pregnancy.

Interventions: For the prospective component eligible patients will be consented and enrolled. A vancomycin trough level will be determined as normal standard of care thirty minutes prior to the appropriate vancomycin dose, followed by a vancomycin peak level one hour after the end of the infusion. Serum concentration time data will then be used to calculate an AUC. The retrospective component of the study will involve a chart review of patients treated with vancomycin in which a serum trough and peak level was obtained and calculation of the AUC as described.

Evaluations: Serum concentration time data will be used to calculate an AUC for each patient enrolled in the study and from all charts reviewed that meet criteria. MIC data will be determined for Staphylococcus aureus isolates obtained from The Nebraska Medical Center. The two sets of data will then be used to calculate an AUC:MIC ratio. The AUC:MIC data will be compared to the goal ratio of greater than 400. Additionally, using the AUC data from our patients and the MICs derived from a large national surveillance data base, a Monte Carlo analysis will be completed to determine the probability of achieving therapeutic ratios.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Admitted to an inpatient care unit at The Nebraska Medical Center
* Prescribed intravenous vancomycin therapy with a dosing interval of 24 hours or less
* Vancomycin therapy that lasts for at least 3 doses or 5 half-lives as scheduled with no dosage changes

Exclusion Criteria:

* Estimated creatinine clearance (CrCl) less than 30 ml/min using the Cockroft-Gault equation (in patients over the age of 65 a SCr of 1.0 mg/dL will be assumed for all patients with a reported SCr less than 1.0 mg/dL). Ideal body weight will be used for the Cockroft-Gault equation unless the actual body weight is less than the ideal body weight.
* Patients requiring any form of dialysis
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected or documentd staphylcoccus aureus infection and prescribed vancomycin
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2011-02-03 (Actual); Study Completion 2011-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of vancomycin dosing regimens achieving AUC:MIC ratio > 400 | 12 months
  The primary outcome is the percentage of vancomycin dosing regimens that achieve AUC:MIC ratio > 400 on the first occurrence of vancomycin use in patients with a suspected or documented S. aureus infection at The Nebraska Medical Center.

SECONDARY OUTCOMES:
Therapeutic vancomycin threshold | 12 months
  Using MIC data from the TRUST Study database and the vancomycin AUC data obtained from TNMC patients, perform a Monte Carlo analysis that will assess the probability of achieving a therapeutic vancomycin threshold with a large number of isolates

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Olsen, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States